CLINICAL TRIAL: NCT04709939
Title: Determining the Acceptability and Feasibility of Mobile-health Approaches to Gather Clinical Information From Patients at Home Following Hospital Discharge
Brief Title: Mobile-health Approach to Gather Clinical Information From Patients Following Hospital Discharge
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Philip Polgreen, Professor, Internal Medicine, University of Iowa
Other Study IDs: 202010084; R21TR003410 (NIH)
Record Dates: First submitted 2020-12-11; First posted 2021-01-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Outpatient Parenteral Antibiotic Therapy
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Participants: Adults patients who are discharged from the hospital on outpatient parenteral antibiotic therapy.
  Interventions: Other: OPAT
- Physician Participants: Infectious disease physicians who prescribe OPAT to their patients but were not involved in the study.
  Interventions: Other: Focus Group

INTERVENTIONS:
Other: OPAT — Observation of patients who are discharged from the hospital on OPAT.
  Groups: Patient Participants
Other: Focus Group — Focus group with infectious disease physicians who prescribe OPAT to patients but were not involved in the study.
  Groups: Physician Participants

SUMMARY:
The purpose of this study is to assess the feasibility of using a mobile-health approach to gather clinical data from patients following discharge from the hospital on outpatient parenteral antibiotic therapy (OPAT). The study population will consist of adult participants who have a smartphone that is capable of both text messaging and pairing with a Bluetooth thermometer that will be provided. Following discharge, patients will be asked to respond to two daily text messages. They will also be reminded to take and send in photos of any skin rashes that may develop as well as their PICC-line site during dressing changes. Text messages will be sent for up to 30 days, but will be stopped sooner if the patient is readmitted to the hospital or if OPAT is discontinued. At the end of the 30 days, all patients will be sent a text message survey about usability, the time it took to complete the study tasks, suggestions for future improvements, and whether they would be willing to be interviewed via phone. A subset of the participants will be interviewed via phone to obtain more detailed feasibility data. Information from the patient's medical record will be collected at the time of hospital discharge as well as at the end of the study period.

Additionally, a focus group (via conference call) will be conducted with all research team members and infectious disease physicians involved in OPAT who did not use the system to gauge their needs and to get ideas for future applications of our tools.

DETAILED DESCRIPTION:
Following hospital discharge on OPAT, patients will be asked to respond to two daily text messages, one in the morning and one in the evening. The message will 1) ask them to take their temperature using the provided thermometer, 2) will provide a link to a web-based survey that will ask about any symptoms as well as provide a free text response field, and 3) remind them to take and send in any photos of any skin rashes that may develop as well as their PICC-line site during dressing changes. Text messages will be sent for up to 30 days, but will be stopped sooner if the patient is readmitted to the hospital or if OPAT is discontinued. At the end of the 30 days, all patients will be sent a text message survey about usability, the time it took to complete the study tasks, suggestions for future improvements, and whether they would be willing to be interviewed via phone. A subset of the participants will be interviewed via phone to obtain more detailed feasibility data.

Additional information will also be collected from the patient and their medical record at the time of hospital discharge (patient caregiver situation, pronouns to address them, artificial material in joints or bones, biological sex, race, ethnicity, height, weight, BMI, zip code, insurance, reason for OPAT, organisms in cultures, where patient is receiving discharge medication, discharge medications, and any other diagnoses/co-morbidities) as well as 2 months after enrollment (any readmission dates and reasons, emergency room visit dates and reasons, clinic visit dates and reasons, and medication changes within 30 days of starting OPAT). These data will be collected 2 months after enrollment to ensure that all readmissions, visits, and medication changes are captured in the medical record.

The software will save time-stamped responses to all web-based surveys, photos sent in, and temperatures taken by the thermometer.

Additionally, a focus group will be conducted (via conference call) with all research team members and infectious disease physicians involved in OPAT who did not use the system to gauge their needs and to get ideas for future applications of our tools. This conference call will be video and audio recorded.

There will not be any long-term follow up for the study.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 18 to 100
* Being discharged from hospital on OPAT
* Owns a smartphone capable of text messaging and being paired to Bluetooth thermometer
* Able to send SMS and MMS messages via phone

Patient Exclusion Criteria:

* Prisoner status
* Unable to provide own written, informed consent

Physician Inclusion Criteria:

* Infectious disease physician who prescribes OPAT

Physician Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being discharged from hospital on OPAT.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-11-19 (Actual)

PRIMARY OUTCOMES:
Number of Days with a Temperature Reading | 30 days
  The number of days that participants submit a temperature reading during the course of the study.
Number of Completed Surveys | 30 days
  The number of completed surveys that the participant submits over the course of the study.
Number of Photos Sent | 30 days
  The number of photos that the participant submits over the course of the study.
Sample Size Estimation for Future Study | 30 days
  The sample size required to conduct a powered study in the future.

SECONDARY OUTCOMES:
Suggestions for Future Use survey | 30 days
  Feedback from focus group participants for future applications of the methods.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Polgreen, MD, MPH, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No